CLINICAL TRIAL: NCT01918488
Title: Increased Activity of the Epithelial Sodium Channel (ENaC) in Diabetic Nephropathy
Brief Title: Increased Activity of a Renal Salt Transporter (ENaC) in Diabetic Kidney Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); Region of Southern Denmark (Other); The Ministry of Science, Technology and Innovation, Denmark (Other Government); Danish Heart Foundation (Other)
Responsible Party: Principal Investigator, Henrik Andersen, MD, MD, PhD student, University of Southern Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2013-052; 13-04-R94-A4513-22770 (Other Grant/Funding Number: The Danish Heart Foundation)
Record Dates: First submitted 2013-07-31; First posted 2013-08-07 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Diabetic Nephropathies; Hypertension
Keywords: Diabetic Nephropathies; Hypertension; Proteinuria; Albuminuria; Epithelial Sodium Channels; Epithelial Sodium Channel Blockers; Amiloride
MeSH Terms: conditions — Diabetic Nephropathies; Hypertension; Proteinuria; Albuminuria | interventions — Amiloride; Triamterene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nephropathy (Experimental): Diabetics with diabetic nephropathy receiving first a standardized salt diet (200 mmol NaCl/day) for 4 days and then amiloride tablet 20 mg two times daily (morning and afternoon) for 2 days.
  Interventions: Dietary Supplement: Standardized salt diet; Drug: Amiloride
- Control (Experimental): Diabetics without nephropathy receiving a standardized salt diet (200 mmol NaCl/day) for 4 days, then amiloride tablet 20 mg two times daily (morning and afternoon) for 2 days.
  Interventions: Dietary Supplement: Standardized salt diet; Drug: Amiloride

INTERVENTIONS:
Dietary Supplement: Standardized salt diet — 200 mmol NaCl per day given as three meals daily for 4 consecutive days.
Drug: Amiloride — Amiloride tablet 20 mg two times daily (morning and afternoon) for two consecutive days.
  Other Names: Triamterene

SUMMARY:
The purpose of the study is to determine whether a diuretic drug called amiloride is capable of increasing renal salt excretion and thereby decrease blood pressure in diabetic patients with kidney disease. Our hypothesis states that amiloride is capable of reducing blood pressure in these patients and thus decrease the cardiovascular risk associated with diabetic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Negative pregnancy test at inclusion and taking contraceptive medication
* One group with diabetic nephropathy and overt proteinuria
* One normoalbuminuric group without nephropathy
* Creatinine clearance > 40 ml/min

Exclusion Criteria:

* Type 2 diabetes
* Receiving amiloride, glucocorticoids, aldosterone or spironolactone
* Clinically relevant organic or systemic disease including malignancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
24-hour urinary sodium excretion induced by amiloride | Change from baseline urinary sodium excretion at 24 hours after amiloride administration

SECONDARY OUTCOMES:
Office blood pressure measurements | Change from baseline office blood pressure at day 4 of salt diet and at 24 hours after amiloride administration

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Andersen, MD, Principal Investigator — University of Southern Denmark; Jan Erik Henriksen, MD, PhD, Study Director — Odense University Hospital; Claus Bistrup, MD, PhD, Study Director — Odense University Hospital; Boye L Jensen, MD, PhD, Study Director — University of Southern Denmark
Locations (1):
- Cardiovascular and Renal Research, Odense, Denmark

REFERENCES:
- [Background] Svenningsen P, Bistrup C, Friis UG, Bertog M, Haerteis S, Krueger B, Stubbe J, Jensen ON, Thiesson HC, Uhrenholt TR, Jespersen B, Jensen BL, Korbmacher C, Skott O. Plasmin in nephrotic urine activates the epithelial sodium channel. J Am Soc Nephrol. 2009 Feb;20(2):299-310. doi: 10.1681/ASN.2008040364. Epub 2008 Dec 10. PMID 19073825
- [Background] Svenningsen P, Uhrenholt TR, Palarasah Y, Skjodt K, Jensen BL, Skott O. Prostasin-dependent activation of epithelial Na+ channels by low plasmin concentrations. Am J Physiol Regul Integr Comp Physiol. 2009 Dec;297(6):R1733-41. doi: 10.1152/ajpregu.00321.2009. Epub 2009 Sep 30. PMID 19793956
- [Background] Saha C, Eckert GJ, Ambrosius WT, Chun TY, Wagner MA, Zhao Q, Pratt JH. Improvement in blood pressure with inhibition of the epithelial sodium channel in blacks with hypertension. Hypertension. 2005 Sep;46(3):481-7. doi: 10.1161/01.HYP.0000179582.42830.1d. Epub 2005 Aug 22. PMID 16116042
- [Background] Buhl KB, Friis UG, Svenningsen P, Gulaveerasingam A, Ovesen P, Frederiksen-Moller B, Jespersen B, Bistrup C, Jensen BL. Urinary plasmin activates collecting duct ENaC current in preeclampsia. Hypertension. 2012 Nov;60(5):1346-51. doi: 10.1161/HYPERTENSIONAHA.112.198879. Epub 2012 Sep 17. PMID 22987920
- [Derived] Isaksson GL, Hinrichs GR, Andersen H, Bach ML, Weyer K, Zachar R, Henriksen JE, Madsen K, Lund IK, Mollet G, Bistrup C, Birn H, Jensen BL, Palarasah Y. Amiloride Reduces Urokinase/Plasminogen-Driven Intratubular Complement Activation in Glomerular Proteinuria. J Am Soc Nephrol. 2024 Apr 1;35(4):410-425. doi: 10.1681/ASN.0000000000000312. Epub 2024 Jan 23. PMID 38254266